CLINICAL TRIAL: NCT04941209
Title: imPulse™ Una Infrasound-to-ultrasound E-stethoscope 2-minute to Result COVID-19 Self-directed & Point-of-care Screening Test
Brief Title: imPulse™ Una Infrasound-to-ultrasound E-stethoscope
Status: Completed | Type: Observational
Sponsor: Level 42 AI, Inc. (Industry)
Collaborators: Asian Institute of Public Health (Other); Institut de Recherche en Santé de Surveillance Epidemiologique et de Formation (IRESSEF) (Unknown); Laboratoire de la foundation Gombes (Unknown)
Responsible Party: Sponsor
Other Study IDs: L42AI-20210003
Record Dates: First submitted 2021-06-20; First posted 2021-06-28 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Covid19; COVID-19 Pneumonia; COVID-19 Respiratory Infection; COVID-19 Acute Respiratory Distress Syndrome; Mass Screening; Corona Virus Infection; Vaccine Virus Shedding
Keywords: infrasound; ultrasound; vibroacoustics; vibrome; digital-biosignature; e-stethoscope
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — COVID-19 Nucleic Acid Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Inpatients/Outpatients with confirmed COVID-19 with and without pulmonary symptoms.
  Interventions: Device: imPulse™ Una infrasound-to-ultrasound e-stethoscope; Diagnostic Test: (PPA >95%) FDA EUA RT-PCR; Radiation: HR-CT-scan
- Matched-Control: Outpatients without COVID-19 without known non-pulmonary diagnoses or symptoms.
  Interventions: Device: imPulse™ Una infrasound-to-ultrasound e-stethoscope; Diagnostic Test: (PPA >95%) FDA EUA RT-PCR

INTERVENTIONS:
Device: imPulse™ Una infrasound-to-ultrasound e-stethoscope — The imPulse™ System is an every/anywhere-point-of-care cardiopulmonary functional state assessment platform designed to capture normal and abnormal, audible and inaudible cardiopulmonary sounds, rhythms and patterns, via a real-time, intelligent, full-spectrum phonocardiogram obtained from direct to skin coupling or through a layer of clothing.
Diagnostic Test: (PPA >95%) FDA EUA RT-PCR — Real-time RT-PCR that detects amplified SARS-CoV-2 genome in sputum, nasopharyngeal or oropharyngeal swabs, bronchoalveolar lavage fluid, nasal or nasopharyngeal aspirate, and lower respiratory tract aspirates.
  Other Names: RT-PCR
Radiation: HR-CT-scan — High-resolution computer tomography, or CT/CAT, is an X-ray scan that produces images of the chest and is used as a confirmatory test in symptomatic patients that have a negative PCR test.
  Other Names: CT; CAT
  Groups: Case

SUMMARY:
This study generates robust, uniform clinical data across emerging COVID-19 strains to train ML/AI algorithms of the Sponsor's imPulse™ Una infrasound-to-ultrasound e-stethoscope for digital diagnostic feature synthesis of asymptomatic and symptomatic COVID-19 digital biosignatures for rapid and accurate adult and child mass screening.

DETAILED DESCRIPTION:
For the next few years or more, the planet probably won't have enough vaccine for everyone. Even as countries with large COVID-19 vaccination programs start pushing to resume travel and trade:

We will not know who is vaccinated and who is not . We will not know who is an (a)symptomatic COVID-19 carrier and who is not.

Because of this, the global community will remain in various stages of masking, social distancing, lock-down, and limited congregation because of cyclical COVID-19 spikes and people will continue to feel unsafe and afraid as novel COVID-19 variants appear and disappear.

This large-scale, multi-site, multi-national study is informed by a completed pilot study at Johns Hopkins- NCT04556149. This study is designed to validate the ability of the imPulse™ Una infrasound-to-ultrasound e-stethoscope to rapidly and accurately screen outpatients with and without confirmed COVID-19 with sensitivity, specificity, positive and negative predictive value matching (PPA >95%) for early, accurate, and rapid, self-directed and point-of-care diagnosis of COVID-19 in areas still lagging in access to vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and willingness to comply with study procedures
* Inpatient Cases - hospitalized patients with positive COVID-19 PCR test, collected from a respiratory sample within the last 7 days, AND pulmonary symptoms within 72 hours of enrollment
* Outpatient Cases - participant being screened for COVID-19 with positive COVID-19 PCR test respiratory sample Controls - Outpatients with negative COVID-19 PCR test respiratory sample and no pulmonary diagnosis or symptoms Cases or Control not able to sit or stand will be allowed to participate in just the parts of the staircase exam they're capable of doing.

Exclusion Criteria:

* Assisted ventilation, including high flow nasal cannula, or ventilator support
* Unable to comply with study procedures, defined at investigator's discretion
* Participants with any visible skin infections or open wounds in areas where the imPulse™ Una device would be applied

Min Age: 6 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Women/girls and men/boys meeting enrollment criteria will be recruited from among hospitalized inpatients and outpatients with asymptomatic and symptomatic COVID-19 infection. One outpatient control without lung disease or pulmonary symptoms will be selected for each enrolled case.
Sampling Method: Probability Sample
Enrollment: 702 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Digital vibroacoustic biomarker diagnostic performance characteristics | Enrollment through to study completion (min 48hrs through to 3 months)
  Sensitivity, specificity, positive and negative predictive values - of the imPulse™ Una device for point-of-care diagnosis of COVID-19.

SECONDARY OUTCOMES:
imPulse™ Una infrasound-to-ultrasound e-stethoscope device safety | Enrollment through to study completion (min 48hrs through to 3 months)
  Device safety

CONTACTS AND LOCATIONS:
Locations (3):
- Laboratoire de la foundation Gombes, Pointe Noire, Kouilou, Democratic Republic of the Congo
- Asian Institute of Public Health, Bhubaneswar, Odisha, India
- Institute for Health Research, Epidemiological Surveillance and Training ( IRESSEF), Dakar, Almadies, Senegal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: SARS-CoV-2/COVID-19 Study of the Audible and Inaudible Vibroacoustic E-stethoscope - imPulse™ Una — https://clinicaltrials.gov/ct2/show/study/NCT04556149?term=infrasound&draw=2